CLINICAL TRIAL: NCT00005540
Title: Physical Fitness and Cardiovascular Mortality in Firefighters
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Wendy Mack, Professor, University of Southern California
Other Study IDs: 5080; R01HL058227 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study prospectively the interrelationships among physical fitness, activity, other measured risk factors, coronary heart disease (CHD) and all-cause mortality in a cohort of 3,403 firefighters.

DETAILED DESCRIPTION:
BACKGROUND:

From 1971-1991 the Occupational Health Service of Los Angeles Country measured physical fitness and other CHD risk factors (including physical activity, anthropometric measures, blood pressure, smoking, family history of CHD, and levels of total cholesterol, uric acid, and glucose) in Los Angeles County firefighters at application and routine intervals (approximately every three years). The entire cohort of 3403 firefighters is now followed for mortality up to 1996.

DESIGN NARRATIVE:

The entire cohort of 3,403 firefighers is followed up to 1996 in this longitudinal study. The investigators are using a variety of tracing sources, including the National Death Index, and obtaining death certificates to determine date and cause of death. Cohort data will be analyzed to address the following aims: (1) To provide a longitudinal description of and determine the interrelationships among physical fitness, physical activity, and other measured risk factors; (2) to determine whether levels of physical fitness are related, independently of other known and measured risk factors, CHD and all-cause mortality; (3) To determine whether there is a gradient of decreasing CHD risk with increasing levels of physical fitness, or whether there appears to be some threshold of physical fitness, above which CHD risk stabilizes; (4) To determine whether the relationship between physical fitness and CHD and all-cause mortality varies by such cardiovascular risk factors as age, cholesterol levels, blood pressure, smoking, and obesity.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3403 (Actual)
Dates: Start 1999-07; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Mack — University of Southern California

IPD SHARING:
Plan to Share IPD: No